CLINICAL TRIAL: NCT04152512
Title: Quality of Life, Specific Needs and Satisfaction With Care After Treatment for Vulvar Cancer - a Prospective, Longitudinal Swedish Nationwide Study
Brief Title: Quality of Life, Unmet Needs and Satisfaction With Care After Vulvar Cancer
Acronym: PROVE
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Diana Zach, MD, senior consultant, Karolinska University Hospital
Other Study IDs: 2018/1402-31/1
Record Dates: First submitted 2019-10-27; First posted 2019-11-05 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Vulvar Cancer; Quality of Life
Keywords: Questionnaire; EORTC QLQ C30 + VU34; Hospital Depression and Anxiety Scale; EORTC-PATSAT; Supportive Care Needs Survey Short Form
MeSH Terms: conditions — Vulvar Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole Cohort: Whole cohort administration of questionnaire at 7 times
  Interventions: Behavioral: Questionnaire administration

INTERVENTIONS:
Behavioral: Questionnaire administration — Questionnaire administration (4 different forms: pre-treatment, 3-4 months after treatment, 1 year after treatment, 2-5 years (yearly) after treatment

SUMMARY:
The aim of this prospective, longitudinal Swedish multi-center study is to assess the quality of life, treatment-related morbidity, unmet needs and satisfaction with care after treatment for vulvar cancer, evaluated by a validated questionnaire.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Information about:

* General and vulvar-cancer-specific quality of life before and after any treatment for newly diagnosed vulvar cancer
* Treatment-related morbidity after any treatment for newly diagnosed vulvar cancer
* Unmet needs of patients with newly diagnosed vulvar cancer
* Satisfaction with care after any treatment for newly diagnosed vulvar cancer in Sweden.

OUTLINE:

The study is planned as a prospective, longitudinal multi-centre study in Sweden. Since 2017, the treatment of vulvar cancer patients has been accredited to four tertiary referral university hospitals in Sweden; the Sahlgrenska University hospital in Gothenburg, the Linköping University hospital, the Skåne University hospital in Lund and the Karolinska University hospital in Stockholm.

150 patients are estimated for inclusion during a time frame of about 18 months.

Eligible patients will be asked to complete a validated questionnaire at different points of time (before and after treatment). Calculating a response rate of about 50% - 60%, this will result in at least 80 completed questionnaires.

The questionnaires consist of the following parts:

* European Organisation for Research and Treatment of Cancer (EORTC)-QLQ-C30
* European Organisation for Research and Treatment of Cancer (EORTC)-QLQ-VU-34 (Vulva-specific module)
* Hospital Depression and Anxiety Scale (HADS)
* Supportive Care Needs Survey Short Form, excerpt (SCNS-SF34)
* European Organisation for Research and Treatment of Cancer (EORTC)-PATSAT (Patient Satisfaction), excerpt
* Demographic data
* 25 self-constructed (and validated) questions

RESULTS:

Results are expected to be available in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of vulvar cancer, all stages, all planned treatments
* Informed consent

Exclusion Criteria:

* Disability to understand and complete the questionnaire due to language difficulties, severe psychiatric illness or dementia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed invasive vulvar cancer in Sweden during the study time frame.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Global quality of life | 1 year after end of treatment
  Measured by the European Organisation of Research and Treatment of Cancer (EORTC)-QLQ-C30-questionnaire.
  Measurement on a scale between 0-and 100. Higher values represent better quality of life. A change of at least 5-8 points is regarded as clinically significant.
Vulvar-cancer-specific quality of life | 1 year after end of treatment
  Measured by the EORTC-QLQ-VU34-questionnaire. Higher values represent higher quality of life.

SECONDARY OUTCOMES:
Satisfaction with Care | 3--4 months after end of treatment
  Measured by EORTC-PATSAT-questionnaire. Higher score represent higher satisfaction with care.
Depression and anxiety | 1 year after end of treatment.
  Measured by the Hospital Anxiety and Depression Index (HADS)-questionnaire. Higher scores represent more depression and anxiety
Unmet needs | 3-4 months after end of treatment.
  Measured by the Supportive Care Needs Survey-Short Form (SCNS-SF)-34-questionnaire. Higher scores represent higher needs.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Zach, MD, Principal Investigator — Karolinska University Hospital, Karolinska Institute, Stockholm, Sweden
Locations (4):
- Sweden (4):
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg
  - Linkopings University Hospital, Linköping
  - Skanes University Hospital Lund, Lund

REFERENCES:
- [Derived] Zach D, Jensen PT, Falconer H, Kolkova Z, Bohlin KS, Kjolhede P, Raices Cruz I, Avall-Lundqvist E, Floter Radestad A. The impact of local symptoms on health-related quality of life in vulvar cancer survivors-A nationwide prospective study. Acta Obstet Gynecol Scand. 2025 Aug;104(8):1517-1529. doi: 10.1111/aogs.15164. Epub 2025 Jun 9. PMID 40490985